CLINICAL TRIAL: NCT02468726
Title: A Clinical Investigation to Demonstrate the Performance of NER1008 Enema in Bowel Cleansing Compared to Fleet® Enema
Brief Title: Performance of NER1008 Enema Compared With Fleet® Enema in Bowel Cleansing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: NER1008-01/2011 (ENE)
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2011-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- NER1008 (Experimental): Use of NER1008 enema for bowel cleansing
  Interventions: Device: NER1008 enema
- Fleet (Active Comparator): Use of Fleet enema for bowel cleansing
  Interventions: Drug: Fleet

INTERVENTIONS:
Device: NER1008 enema — NER1008 enema administered to cleanse the bowel bewteen 1 and 3 hours prior to flexible sigmoidoscopy
  Arms: NER1008
Drug: Fleet — Fleet enema administered to cleanse the bowel bewteen 1 and 3 hours prior to flexible sigmoidoscopy
  Arms: Fleet

SUMMARY:
In order for flexible sigmoidoscopy to be a successful screening procedure, the bowel must be free of solid matter so the endoscopist has a clear view, increasing the chance of detection of abnormalities. This is achieved through the use of bowel cleansing preparations, which are administered prior to the procedure. Enemas are the preferred method as they clear the lower bowel more quickly than oral formulations and do not require dietary restrictions.

The medical device being tested in this clinical investigation is NER1008, an enema which contains PEG3350 (polyethylene glycol 3350). PEG3350 is an osmotic agent, which holds the water content in the rectum and sigmoid colon, consequently increasing stool volume, resulting in rectal distension and subsequent distal colon emptying. The increased colonic luminal content stimulates the motility, propulsive transportation and rectal evacuation of the distal colon content.

This study is designed to assess the performance of NER1008 in bowel cleansing and compare this with the performance of Fleet® enema, which is widely used for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects [as determined by medical history, physical examination, laboratory test values, vital signs and 12-lead electrocardiograms (ECG's) at screening] aged 18 to 45 years.
2. Non-smokers from 3 months before enema administration and for the duration of the clinical investigation.
3. Body mass index (BMI) ≥ 18 and ≤ 35 kg/m2.
4. Must voluntarily provide written informed consent to participate in the clinical investigation.
5. Must understand the purposes and risks of the clinical investigation and agree to follow the restrictions and schedule of procedures as defined in the clinical investigation plan, and as confirmed during the informed consent process.
6. Female subjects must be postmenopausal (for at least one year and confirmed by a serum follicle stimulating hormone (FSH) test at screening), surgically sterile, practising true sexual abstinence or must use an effective method of contraception.
7. Female subjects of child-bearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at check-in of each period.
8. The subject's primary care physician must confirm that there is nothing in their medical history that would preclude their enrolment into this clinical investigation.
9. Must be willing to consent to have data entered into The Over Volunteering Prevention System (TOPS).

Exclusion Criteria:

1. Subjects with a history or presence of significant cardiovascular disease, pulmonary, hepatic, gallbladder or biliary tract, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.
2. Subjects with a history or presence of organic or functional gastrointestinal conditions (e.g. chronic constipation, irritable bowel syndrome, inflammatory bowel disease).
3. Subjects with a clinically relevant history or presence of abnormal gastrointestinal motility.
4. Subjects with a significant history of hereditary bowel disorders.
5. Subjects with abnormal findings on the digital rectal examination performed at screening.
6. Use of laxatives or motility altering drugs in the 3 months preceding enema administration.
7. Use of any prescription or over-the-counter medication (including vitamins, herbal and mineral supplements) within 14 days prior to enema administration (or within 5 half lives if longer), with the exception of Investigator-approved hormonal contraceptives, hormone replacement therapy (HRT) and occasional paracetamol.
8. Participation in a clinical drug study during the 30 days preceding enema administration in this clinical investigation.
9. Donation of blood or blood products within 30 days prior to enema administration or during the clinical investigation, except as required for this clinical investigation
10. Pregnant or lactating females.
11. Any clinically significant illness within 28 days prior to enema administration.
12. History or presence of any significant drug allergy, or a known allergy or contraindication to polyethylene glycols, Fleet® enema or midazolam.
13. Laboratory values at screening which are deemed to be clinically significant, unless agreed in advance by the Sponsor's Medical Representative and Principal Investigator.
14. Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
15. Current or history of drug or alcohol abuse within the 12 months prior to enema administration, or a positive drugs of abuse test at screening or check-in.
16. Consumption of alcoholic beverages within 24 hours of confinement or during confinement.
17. Subjects who, in the opinion of the Investigator, are unsuitable for participation in the clinical investigation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Success of bowel cleansing | Up to 3 hours
  Whether recto-sigmoid bowel cleansing has been successful, based on an endoscopist's assessment of the quality of cleansing in the rectum and colon, according to the modified Harefield cleansing scale.

SECONDARY OUTCOMES:
Grade of bowel cleansing | Up to 3 hours
  Grade of bowel cleansing (A, B, C or D), based on an endoscopist's assessment.
Quality of cleansing in rectum | Up to 3 hours
  Quality of cleansing in the rectum based on the modified Harefield cleansing scale (0-4).
Quality of cleansing in sigmoid colon | Up to 3 hours
  Quality of cleansing in the sigmoid colon based on the modified Harefield cleansing scale (0-4)
Quality of cleansing in the descending colon | Up to 3 hours
  Quality of cleansing in the descending colon to the splenic flexure based on the modified Harefield cleansing scale (0-4)
Depth of scope progression | Up to 3 hours
  Prior to removing the endoscope, the depth of progression it has made, in cms
Stool weight | Up to 3 hours
  Weight of stool during the one hour period after the administration of the enema

CONTACTS AND LOCATIONS:
Overall Officials: David J Bell, MD, Principal Investigator — BioKinetic Europe Ltd
Locations (1):
- BioKinetic Europe Ltd, Belfast, United Kingdom